CLINICAL TRIAL: NCT03651791
Title: In Vivo MRI Tracking of Mesenchymal Stromal Cells Labeled With Ultra-Small Paramagnetic Iron Oxide Particles After Intramyocardial Transplantation in Patients With Chronic Ischemic Heart Disease
Brief Title: In Vivo Tracking of USPIO Labeled MSC in the Heart
Acronym: USPIO-MSC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Bruun Mathiasen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USPIO-MSC1
Record Dates: First submitted 2018-08-23; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- USPIO labeled MSC injection (Experimental): USPIO labeled MSC injection
  Interventions: Combination Product: USPIO labeled MSC injection

INTERVENTIONS:
Combination Product: USPIO labeled MSC injection — USPIO labeled MSC injection

SUMMARY:
To evaluate the ability to trace iron oxide-labeled mesenchymal stromal cells with magnetic resonance imaging (MRI) after NOGA-guided injection therapy into the myocardium in patients with ischemic heart disease.

DETAILED DESCRIPTION:
Aims:

To evaluate the ability to trace iron oxide-labeled mesenchymal stromal cells with magnetic resonance imaging (MRI) after NOGA-guided injection therapy into the myocardium.

To evaluate the safety and efficacy of treatment with iron oxide-labeled mesenchymal stromal cells to form new heart muscle cells and blood vessels in the myocardium submitted by NOGA-guided injection therapy in the myocardium in order to improve myocardial blood flow and reduce patients' symptoms.

Patient Population:

Patients with coronary artery disease not treatable with additional bypass surgery or percutaneous coronary intervention who have angina pectoris (Canadian Cardiovascular Society (CCS) class II-III) or angina equivalent shortness of breath (New York Heart Association (NYHA) class II -III).

Study Design A prospective, non-randomized, pilot study including 5-10 patients. Patients will by means of the percutaneous NOGA injection catheter system receive 12-15 intramyocardial injections. The number depending on the amount of cultured cells and distributed uniformly in the peripheral zone of a presumed ischemic area in the left ventricle demonstrated by angiography, magnetic resonance imaging and NOGA mapping.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 80 years.
* Signed informed consent.
* Chronic stable ischemic heart disease
* New York Heart Association (NYHA) class II-IV or Canadian Cardiovascular Society (CCS) class II-IV
* Maximal tolerable angina and/or heart failure medication.
* Angiography within 12 months of inclusion. Angiography must have at least one larger coronary vessel with a significant stenosis with no option for revascularization (Angiographies evaluated by an independent thoracic surgeon and an interventional cardiologist).
* Patients who have had revascularization done within 6 months of inclusion must have a new angiography at least 4 months after the intervention to rule out early restenosis.

Exclusion Criteria:

* Pregnant or fertile women.
* Clinical significant anemia, leukopenia, leukocytosis or thrombocythemia.
* Diminished functional capacity for other reasons such as: chronic obstructive pulmonary disease (COLD) with Forced Expiratory Volume in 1 second (FEV1)<1 L/min, moderate to severe claudication or morbid obesity.
* Patients with reduced immune response or treated with immunosuppressive medication.
* Moderate to severe valvular disease or valvular disease with option for valvular surgery.
* Acute coronary syndrome with elevation of coronary markers, stroke or Transitory Cerebral Ischemia (TCI) within 6 weeks of inclusion.
* History with malignant disease within 5 years of inclusion or suspected malignity.
* Other experimental treatment within 4 weeks of baseline evaluation.
* Other revascularization treatment within 4 months of treatment.
* Contraindications for Magnetic Resonance Imaging (MRI) such as: Claustrophobia, pacemaker, Implantable Cardioverter Defibrillator (ICD) unit, metal fragments or metal implants in the cranium

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
MSC identification using MRI in-vivo on day 0 | 24 hours
  Being able to identify the iron-oxide labeled mesenchymal stromal cells on day 0 after injection into the myocardium by MRI.

SECONDARY OUTCOMES:
MSC identification using MRI in-vivo on day 1 | 1 day
  Being able to identify the iron-oxide labeled mesenchymal stromal cells on day 1
MSC identification using MRI in-vivo on day 7 | 7 days
  Being able to identify the iron-oxide labeled mesenchymal stromal cells on day 7
MSC identification using MRI in-vivo after 2 weeks | 2 weeks
  Being able to identify the iron-oxide labeled mesenchymal stromal cells after 2 weeks
MSC identification using MRI in-vivo after 4 weeks | 4 weeks
  Being able to identify the iron-oxide labeled mesenchymal stromal cells after 4 weeks
MSC identification using MRI in-vivo after 8 weeks | 8 weeks
  Being able to identify the iron-oxide labeled mesenchymal stromal cells after 8 weeks
MSC identification using MRI in-vivo after 12 weeks | 12 weeks
  Being able to identify the iron-oxide labeled mesenchymal stromal cells after 12 weeks
MSC identification using MRI in-vivo after 26 weeks | 26 weeks
  Being able to identify the iron-oxide labeled mesenchymal stromal cells after 26 weeks
Cardiac pump function changes | 12 weeks
  Left ventricular ejection fraction, systolic and diastolic volumes after 12 weeks
Cardiac pump function changes | 26 weeks
  Left ventricular ejection fraction, systolic and diastolic volumes after 26 weeks
CCS class | 12 weeks
  Canadian Cardiovascular Society (CCS) class after 12 weeks
CCS class | 26 weeks
  Canadian Cardiovascular Society (CCS) class after 26 weeks
Seattle Angina Questionnaire | 12 weeks
  Seattle Angina Questionnaire after 12 weeks
Seattle Angina Questionnaire | 26 weeks
  Seattle Angina Questionnaire after 26 weeks
Weekly number of angina attacks | 12 weeks
  Weekly number of angina attacks after 12 weeks
Weekly number of angina attacks | 26 weeks
  Weekly number of angina attacks after 26 weeks
Weekly nitroglycerin consumption | 12 weeks
  Weekly nitroglycerin consumption after 12 weeks
Weekly nitroglycerin consumption | 26 weeks
  Weekly nitroglycerin consumption after 26 weeks
Adverse events | 6 months
  Adverse events registration

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kastrup, MD DMSc, Study Director — The Heart Centre, Rigshospitalet, University of Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mathiasen AB, Hansen L, Friis T, Thomsen C, Bhakoo K, Kastrup J. Optimal labeling dose, labeling time, and magnetic resonance imaging detection limits of ultrasmall superparamagnetic iron-oxide nanoparticle labeled mesenchymal stromal cells. Stem Cells Int. 2013;2013:353105. doi: 10.1155/2013/353105. Epub 2013 Mar 19. PMID 23577035
- [Background] Hansen L, Hansen AB, Mathiasen AB, Ng M, Bhakoo K, Ekblond A, Kastrup J, Friis T. Ultrastructural characterization of mesenchymal stromal cells labeled with ultrasmall superparamagnetic iron-oxide nanoparticles for clinical tracking studies. Scand J Clin Lab Invest. 2014 Aug;74(5):437-46. doi: 10.3109/00365513.2014.900698. Epub 2014 Apr 15. PMID 24734781
- [Derived] Mathiasen AB, Qayyum AA, Jorgensen E, Helqvist S, Ekblond A, Ng M, Bhakoo K, Kastrup J. In Vivo MRI Tracking of Mesenchymal Stromal Cells Labeled with Ultrasmall Paramagnetic Iron Oxide Particles after Intramyocardial Transplantation in Patients with Chronic Ischemic Heart Disease. Stem Cells Int. 2019 Nov 14;2019:2754927. doi: 10.1155/2019/2754927. eCollection 2019. PMID 31814830